CLINICAL TRIAL: NCT04118517
Title: Bioavailability of Essential Amino Acids From the Common Bean (Phaseolus Vulgaris) in Young Healthy Jamaican Adults Consuming a Typical Meal
Brief Title: Quality of Protein From the Common Bean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Asha Violet Badaloo, Professor, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Protein quality; E4.30.31 (Other: The International Atomic Energy Agency)
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Nutrition Deficiency Due to A Particular Kind of Food
Keywords: protein quality, legume

STUDY DESIGN:
Intervention Model Description: The model is based on the concept that if amino acids in protein become labelled with an isotopic tracer within the food matrix, their appearance in the blood gives a measure of their bioavailability following digestion and absorption of the protein; which is independent of other proteins in the food and independent of endogenous body proteins and gut bacterial proteins. Amino acids in the common bean were labelled with deuterium, by adding a bolus dose of deuterium oxide (2H2O) to the irrigation water. Then a dual tracer technique is used to measure the bioavailability of amino acids in the bean. After consuming a diet prepared with the mature bean, comparative tracer appearance in blood of the deuterium labelled amino acids from the bean and amino acids derived from a reference protein labelled within another tracer (U-13C- spirulina) gives a direct measure of bioavailability of the bean amino acids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test meal (Experimental): The study comprises one arm of 12 healthy Jamaican male and female adults with normal body mass inex, aged 20 to 45 years, receiving a test meal containing the common bean that was intrinsically labelled with deuterium .
  Interventions: Other: Using intrinsically labelled bean protein to assess bioavailability of amino acids in healthy adults

INTERVENTIONS:
Other: Using intrinsically labelled bean protein to assess bioavailability of amino acids in healthy adults — The intervention comprises a test meal of intrinsically deuterium labelled stewed common bean with rice. The meal is mixed with a reference protein (Universally labelled 13C-spirulina, 12 mg/kg) and 13C6-Phenylalanine (0.05mg/kg) which is divided into equal mini meals and fed hourly over 8 hours. Protein in the total meal provides 15% of the energy intake with the labelled bean contributing >50% of the protein.
  Other Names: Testing quality of bean protein in a feeding trial

SUMMARY:
Dietary Protein quality is based on digestion of proteins to amino acids and the bioavailability of the amino acids to maintain good health and body function. Currently, digestibility of proteins, which is measured as the difference between protein intake and faecal loss, is underestimated. This is because, in addition to loss from dietary proteins, faecal loss includes additional protein from gut secretions and bacteria residing in the large intestine. The expert committee on protein quality suggested that a minimally invasive accurate method based on Dual Stable Isotope Tracer approach (non-radioactive) could be developed. This method is based on the concept that if amino acids in proteins become labelled with an isotopic tracer within the food matrix, their appearance in the blood gives a measure of bioavailability. The Food and Agriculture Organization (FAO) of the United Nations and the World Health Organization (WHO) are promoting peas and beans to combat poverty, hunger and malnutrition because they are relatively less expensive sources of protein. We hypothesized that digestibility of protein in the common bean and absorption of amino acids is higher than current estimates.

The aim of this proposal is to conduct a study in 12 healthy adults, aged 20 to 45 years, to test a novel method to assess protein quality of the common bean using the isotopic approach. The Scientific Research Council will grow the labelled beans by adding a tracer dose of deuterium to the irrigation water. The beans are prepared a typical Jamaican meal for consumption. The meal is mixed with a labelled reference protein (U-13C-spirulina) which is universally (U) labelled with stable isotope 13-Carbon (13C) to estimate digestibility; and the amino acid, phenylalanine, in which the 6 ring carbon atoms are labelled with 13C (ring-13C6- phenylalanine) to provide an index of amino acids absorption. Before and after consumption of the meal, samples of blood, breath and urine will be taken. These samples and a sample of the diet will be analysed for amino acids composition and deuterium enrichment using mass-spectrometry. The appearance of each labelled essential amino acid in blood from the bean protein will be calculated. The data will provide accurate date on amino acids bioavailability from the common bean that will be useful for dietary guideline for good health.

DETAILED DESCRIPTION:
Humans require certain minimal quantities of the indispensable amino acids (IAA) from dietary proteins to maintain healthy growth and body function (1). These amino acids are not made in the body and must be provided in the diet. Protein quality is about how dietary proteins can satisfy the body's demand for IAA at various stages of life (1,2) to make different body proteins and biomolecules. It is important to public health and has economic considerations with respect to national food policy, world production and trade in proteins. Uncertainty over the quality of diet, specifically with reference to its protein quality, does potentially impact a nation's health, economy, agriculture and nutrient security. International organizations have begun to address these issues Poor dietary quality has a marked negative impact on the sensitive periods of pregnancy (3) and the first two years of life (the first 1000 days). Furthermore, protein quality is related to stunting which is prevalent in may low and middle income countries because adequate protein quality is required for optimum linear growth. Hence, it is likely to have an impact on the WHO Global Nutrition Target 2025 for reducing the prevalence of stunting (low height-for-age) in children under 5 years by 40%. Stunting has been shown to reduce capacity for learning in children, and hence productivity in adults (4). Of importance, also, stunting increases the risk of developing obesity and chronic non-communicable diseases (CNCD), and therefore plays a role in the impact of CNCD on increasing cost to health and the economy especially in developing countries (5). It is clear that to meet dietary requirements of the IAA, accurate assessment of their availability is essential.

The availability of amino acids from protein sources depends on their amino acids composition and digestibility which have been yardsticks used in the assessment of protein quality. The Food and Agriculture Organization (FAO) in 2011 held an International Symposium on Dietary Protein for Human Health where it was recognized that the current measure of protein availability using oro-faecal nitrogen balance underestimate digestibility because colonic metabolism contributing additional nitrogen to dietary nitrogen is not taken into consideration in the stool loss. The committee concluded that a more robust method of assessing protein quality is needed. Whereas oro-ileal balance is a more accurate method of protein digestibility (6,7), it is an expensive and invasive method, and there is insufficient human data.

Following the symposium in 2011, FAO in 2013 convened a expert consultation meeting and released a report , 'Dietary protein quality evaluation in human nutrition', (8) as part of the call from the United Nations to promote sustainable diets and health and influenced by the 2012 WHO technical note on foods for the management of moderate acute malnutrition in children(9) This report was motivated mainly by advances in methods available to measure the quality of nutritional proteins with more accuracy. It was suggested that a minimally invasive method based on Dual Stable Isotope Tracer approach could be developed to accurately assess protein quality. The IAEA held a Consultants' Meeting in October 2013 to discuss stable isotopic methods to measure protein quality in humans, followed by a FAO Expert Working Group Meeting in March 2014 in Bangalore, to specifically define the most appropriate research methodologies to measure protein digestibility and utilization in humans (10).Hence, the International Atomic Energy Agency (IAEA) has established a Co-ordinated Research Project (CRP) with the aim to develop and validate a novel Dual Stable Isotope Tracer method that is minimally invasive to assess protein digestibility and utilization from plant based diets, as they are consumed by vulnerable populations, in regions habitually relying on plant based diets. Generally, the method is based on the concept that if IAA become labeled with isotope within the food matrix, their appearance in the blood gives a measure of bioavailability, which is independent of other proteins in the food and independent of endogenous body proteins. Comparative tracer appearance in blood of labelled test and reference proteins gives a direct measure of digestion and bioavailability of the test protein. Also, when the reference protein is accompanied by a trace quantity of a differently labelled amino acid such as 13C6-phenylalanine, it will provide an index of amino acids absorption following digestion. We have been awarded an IAEA grant as part of the CRP and proposing to conduct studies in healthy human adults to assess the availability of the IAA from intrinsically labelled common bean (Phaseolus vulgaris) which is among the eight species regarded as global priorities by the Consultative Group for International Agricultural Research (CGIAR, 2012) (11) The research Program includes leveraging legumes to combat poverty, hunger, malnutrition and environmental degradation. Our collaborator from the Scientific Research Council will grow the beans. The amino acids in the bean will be labelled with deuterium, by adding a bolus dose of deuterium oxide to the irrigation water. They have successfully produced labelled beans in a pilot study. To accurately measure IAA availability and protein quality in the common bean will be useful to inform dietary choices consistent with good health The main aim of this study is to develop a minimally invasive method to accurately measure protein quality in the common bean to inform dietary choices consistent with good health. We also, aim to establish an absorption index relative to phenylalanine for use in future studies and to assess utilisation of the protein by measuring protein oxidation and urinary amino acids.

Specific aims are:

1. to characterize the bean protein for isotopic enrichment
2. to quantify bean amino acids made available to the body when the bean and a reference protein are consumed by healthy adults, aged 20 to 45 years.
3. to establish an index for amino acids absorption
4. to determine digestible indispensable amino acids scores

ELIGIBILITY:
Inclusion Criteria:

* Age range - 20-45 years
* BMI range- 18.5 - 25 kg/m2
* Male or Female
* No food allergies

Exclusion Criteria:

* History of diabetes
* History of hypertension, any chronic illness
* Acute illness within the last 2 weeks
* Involved in competitive sports
* Altered sleep/ eating schedules
* Weight loss or gain in the past six months
* Pregnancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Digestibility of protein from the common bean | 8h
  Measured by comparing plasma enrichment of each deuterium labelled indispensable amino acid (IAA) from the bean to plasma enrichment of the same 13C- labelled IAA from a highly digestible reference protein (Universally 13C-labelled spirulina)
Absorption index of amino acids | 8h
  Calculated based on the enrichment of free L-[ring-13C6]-phenylalanine in plasma at steady state divided by its enrichment in the meal.
Digestible indispensable amino acids score | 8h
  mg of digestible bean IAA in 1g bean protein/ mg of the same IAA in 1g reference protein

CONTACTS AND LOCATIONS:
Overall Officials: Asha V Badaloo, PhD, Principal Investigator — University of the West Indies, Mona Campus
Locations (1):
- Tropical Metabolism Research Unit, Caribbean Institute for Health Research, University of the West Indies, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Joint WHO/FAO/UNU Expert Consultation. Protein and amino acid requirements in human nutrition. World Health Organ Tech Rep Ser. 2007;(935):1-265, back cover. PMID 18330140
- [Background] Food and Agriculture Organization, Protein quality evaluation. Report of the Joint FAO/WHO Expert Consultation. FAO food and Nutrition paper 5. FAO 1991
- [Background] Duggleby SL, Jackson AA. Relationship of maternal protein turnover and lean body mass during pregnancy and birth length. Clin Sci (Lond). 2001 Jul;101(1):65-72. PMID 11410116
- [Background] Hoddinott J, Maluccio JA, Behrman JR, Flores R, Martorell R. Effect of a nutrition intervention during early childhood on economic productivity in Guatemalan adults. Lancet. 2008 Feb 2;371(9610):411-6. doi: 10.1016/S0140-6736(08)60205-6. PMID 18242415
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Moughan PJ. Amino acid availability: aspects of chemical analysis and bioassay methodology. Nutr Res Rev. 2003 Dec;16(2):127-41. doi: 10.1079/NRR200365. PMID 19087386
- [Background] Fuller MF, Tome D. In vivo determination of amino acid bioavailability in humans and model animals. J AOAC Int. 2005 May-Jun;88(3):923-34. PMID 16001870
- [Background] Dietary protein quality evaluation in human nutrition. Report of an FAQ Expert Consultation. FAO Food Nutr Pap. 2013;92:1-66. No abstract available. PMID 26369006
- [Background] World Health Organization (2012), Technical Note: Supplementary foods for the management of moderate acute malnutrition in infants and children 6-59 months of age, WHO, Geneva.
- [Background] Lee WT, Weisell R, Albert J, Tome D, Kurpad AV, Uauy R. Research Approaches and Methods for Evaluating the Protein Quality of Human Foods Proposed by an FAO Expert Working Group in 2014. J Nutr. 2016 May;146(5):929-32. doi: 10.3945/jn.115.222109. Epub 2016 Apr 6. PMID 27052532
- [Background] CGIAR. 2012. CGIAR Research Program on Grain Legumes Leveraging legumes to combat poverty, hunger, malnutrition and environmental degradation. Consortium of International Agricultural Research Centers, Montpellier.